CLINICAL TRIAL: NCT06463899
Title: Impact of Bilateral Parasternal Infusion of Local Anesthetics in Patients With Respiratory Risk Factors Over the Length of Hospitalization and Morphine Sparing in the Intensive Care Unit After On-pump Coronary Bypass Surgery
Brief Title: Evaluation of the Effectiveness of the Administration of Local Anesthetics Via Two Catheters Placed During Surgery, and Study of the Benefits on Respiratory Function and Therefore on Recovery Time
Acronym: PARALSTER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PO22011
Record Dates: First submitted 2023-08-14; First posted 2024-06-18 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-06

CONDITIONS: Duration of Hospitalization in Intensive Care Unit
Keywords: para-sternal catheters; analgesia; coronary bypass surgery; sternotomy; hospitalization
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WITH catheter (Experimental): A "multi-perforated catheter" arm benefiting from opioid analgesia (Patient controlled Analgesia ((PCA)) morphine (bolus-only mode or morphine titration if PCA not available), nefopam, non-steroidal anti-inflammatory drugs, ketamine, pregabalin and paracetamol associated with analgesia by continuous infusion of local anesthetics (ropivacaine) via two multi-perforated catheters
  Interventions: Procedure: multi-perforated catheter
- WITHOUT catheter (Active Comparator): A "control" arm benefiting from opioid analgesia (PCA morphine in bolus mode alone or morphine titration if PCA not available), nefopam, non-steroidal anti-inflammatory drugs, ketamine, pregabalin and paracetamol.
  Interventions: Procedure: Classic procedure

INTERVENTIONS:
Procedure: multi-perforated catheter — After skin closure, cardiac surgeons place multi-perforated catheters aseptically.
  Arms: WITH catheter
Procedure: Classic procedure — opioid analgesia (PCA morphine in bolus mode alone or morphine titration if PCA not available), nefopam, non-steroidal anti-inflammatory drugs, ketamine, pregabalin and paracetamol
  Arms: WITHOUT catheter

SUMMARY:
Currently intravenous analgesics are used for postoperative analgesia. But the analgesia of these products is tempered by their adverse effects (sedation, confusion, nausea or vomiting, delayed transit, urinary retention and pruritus) which can slow down postoperative recovery.

The aim of this study is to evaluate the effectiveness of the administration of local anesthetics via two catheters placed during surgery, but also to study their benefit on respiratory function and therefore on recovery time and morphine sparing.

DETAILED DESCRIPTION:
Medical context:

Cardiac surgery and more specifically coronary bypass surgery are very painful postoperative surgeries, especially during the first 48 hours following the operation. These pains, present at rest, are increased when the patient is mobilized, during coughing, deep inspiration, chairing or mobilization in bed.

In cardiac surgery, it has been shown that respiratory complications remain a significant cause of morbidity and mortality. They can lead to an extension of the length of hospitalization and therefore an increase in hospital costs. Indeed, these are increased compared to other surgeries because of the sternotomy and the pain it causes, as well as the type of ventilation during extracorporeal circulation (sharp reduction or even stopping of mechanical ventilation).

Patients having, prior to surgery, risk factors for postoperative respiratory complications, present increased risks of pneumonia, postoperative atelectasis, pleurisy, re-intubation, mortality and therefore an additional cost of hospitalization.

Limiting postoperative pain allows better rehabilitation of the patient by improving patient mobilization, participation in respiratory physiotherapy and therefore potentially a reduction in respiratory complications.

Currently, multimodal analgesia combining opioids, nefopam, nonsteroidal anti-inflammatory drugs, ketamine, lidocaine and paracetamol, is the most widely used technique in patients. The analgesic efficacy provided by opioids is tempered by their side effects (sedation, confusion, nausea or vomiting, transit delay, urinary retention, pruritus) which may slow postoperative recovery. In addition, opioids can also decrease the cough reflex and impair respiratory control.

It is therefore important to find alternatives to the analgesic management of these patients who, thanks to the improvement of surgical and anesthetic techniques, are more and more numerous.

The use of para-sternal catheters with bilateral infusion of local anesthetics has already shown its effectiveness in terms of reducing opioid consumption and safety. However, no benefit has yet been proven in terms of reducing the length of hospital stay in subjects at respiratory risk undergoing surgery such as on pump coronary bypass surgery.

Goal :

Show that the use of a bilateral para-sternal infusion of local anesthetics (ropivacaine 0.2%) by multi-perforated catheters in patients with respiratory risk factors who have undergone coronary bypass surgery, makes it possible to reduce the length of stay in an intensive care unit.

ELIGIBILITY:
This study will include adults over 18 years of age requiring on-pump coronary bypass surgery with at least one of the following respiratory risk factors:

* BMI > or = 30 Kg / m2
* Active or withdrawn smoking for less than 6 weeks
* COPD documented by pulmonologist or respiratory function test (LVEF/ FVC <0.7 not reversible after bronchodilator)
* Restrictive ventilatory disorders, defined by a CPT less than 80% of normal
* Chronic respiratory failure, defined by a PaO2, at rest, in ambient air, less than 70 mmHg
* Age > or = 75 years old exclusion criteria:

Any patient meeting one of the following criteria will be excluded from the study:

* Emergency surgery
* Other operative procedure planned during the same intervention (for example vascular), apart from the saphenous sample
* Aortic dissection
* Preoperative renal failure with GFR <30 mL / min / 1.73 m2
* Left heart failure with Ejection fraction <30%
* Pulmonary arterial hypertension> 50 mmHg
* Hepatic cytolysis with ALT or AST> 2N
* ASA score > or = 4
* Coagulopathy
* Anticoagulants or antiaggregants not stopped in time (according to usual protocols) or with poorly performed or unjustified relay
* Chronic use of opioids or history of drug addiction
* Progressive pregnancy or breastfeeding
* Inability to understand protocol and sign consent
* Known allergy to one of the substances in the study protocol
* Patients requiring assistance such as ECMO, intra-aortic counter pulsation balloon or Impella will be excluded from the protocol.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2025-11-08 (Estimated); Study Completion 2026-02-08 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the duration of hospitalization in intensive care unit | Day 1
  Study of the benefit of the administration of local anesthetics via two catheters placed during surgery on recovery time versus currently intravenous analgesics that are used for postoperative analgesia, which are tempered by their adverse effects, and can slow down postoperative recovery.

SECONDARY OUTCOMES:
Evaluation of the pain at rest and on mobilization using a visual pain evaluation scale | Day 2
  Study of the effectiveness of the administration of local anesthetics via two catheters placed during surgery, including their benefit on respiratory function, versus currently intravenous analgesics that are used for postoperative analgesia, which are tempered by their adverse effects.
Evaluation of the total consumption of opioids | At 48 hours
  Study of the use of local anesthetics via two catheters placed during surgery for morphine sparing versus the use of currently intravenous analgesics that are used for postoperative analgesia which are multimodal analgesia combining opioids like nefopam, nonsteroidal anti-inflammatory drugs, ketamine, lidocaine and paracetamol
Evaluation of the patient mortality | Day 30
  Study of the benefit of the administration of local anesthetics via two catheters placed during surgery on respiratory function and complications which remains a significant cause of morbidity and mortality versus currently intravenous analgesics that are used for postoperative analgesia, which are tempered by their adverse effects.
Evaluation of the occurrence of the side effects of opioids | At 48 hours
  Study of the benefit of the administration of local anesthetics via two catheters placed during surgery versus currently intravenous analgesics that are used for postoperative analgesia, which are tempered by their adverse effects as sedation, confusion, nausea or vomiting, delayed transit, urinary retention and pruritus.

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France